CLINICAL TRIAL: NCT01812980
Title: Immunogenicity and Safety of Trivalent Influenza Vaccine in Non-pregnant HIV- Infected Women: An Open Label Trial.
Brief Title: Immunogenicity and Safety of Trivalent Influenza Vaccine in Non-pregnant HIV-infected Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Michelle Groome, Investigator, University of Witwatersrand, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MatFlu_HIVpos_nonpregnant
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Influenza; Human Immunodeficiency Virus
Keywords: Influenza; Human Immunodeficiency Virus
MeSH Terms: conditions — Influenza, Human; Acquired Immunodeficiency Syndrome | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trivalent Inactivated Influenza Vaccine (Experimental): Single dose, intramuscular injection from a pre-filled syringe
  WHO recommendation for influenza vaccines for 2013 for the Southern-hemisphere included the following vaccine strains:
  * an A/California/7/2009 (H1N1)pdm09-like virus;
  * an A/Victoria/361/2011 (H3N2)-like virus; - a B/Wisconsin/1/2010-like virus.
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Inactivated Influenza Vaccine — WHO recommendation for influenza vaccines for 2013 for the Southern-hemisphere included the following vaccine strains:
  * an A/California/7/2009 (H1N1)pdm09-like virus;
  * an A/Victoria/361/2011 (H3N2)-like virus; - a B/Wisconsin/1/2010-like virus.
  Other Names: Vaxigrip

SUMMARY:
The overall aim of this project is to evaluate the immunogenicity of TIV vaccination in HIV-infected non-pregnant women in 2013. Safety data including solicited local and systemic reactions to the vaccine will also be assessed.

DETAILED DESCRIPTION:
Schedule of Events

Visit 1 (enrollment) Informed Consent Form (ICF) signed Inclusion/ exclusion/ Withdrawal criteria Medical history Targeted physical exam Blood draw TIV administered Diary card dispensed

Local/ systematic reactions

Visit 2: 1 month post enrolment (28-35 days) Inclusion/ exclusion/ Withdrawal criteria Medical history Targeted physical exam Blood draw Diary card collected Local/ systematic reactions reviewed

ELIGIBILITY:
Inclusion Criteria:

(i) Documented to be HIV-1 infected on one assay used in the Prevention of Mother to Child Transmission (PMTCT)/ other program undertaken within 12 weeks of study enrolment.

* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of study.
* Not pregnant at time of enrolment (confirmed by urine testing). If pregnant in past year, participant must be at least 6 months post delivery at time of enrolment.
* Women age ≥ 18 years to < 39 years.

Exclusion Criteria:

* Receipt of TIV, other than through the study, during the current and previous two influenza seasons, documented by medical history or record.
* Receipt of any live licensed vaccine ≤ 28 days or any other vaccine (except for tetanus toxoid vaccine) ≤ 14 days prior to study-vaccine.
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) ≤ 28 days prior to vaccination in this study, unless study approval is obtained.
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 38 degrees C ≤ 24 hours prior to study entry.
* Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or has immunosuppression as a result of an underlying illness or treatment.
* Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤ 12 weeks of study entry, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) ≤ 12 weeks before study entry (nasal and topical steroids are allowed).
* Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products.
* Receipt of Interleukin 2, IFN, GMCSF or other immune mediators ≤ 12 weeks before enrollment.
* Uncontrolled major psychiatric disorder.
* History of a severe adverse reaction to previous TIV.
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of Trivalent Influenza Vaccine (TIV)by measuring Hemagglutination Inhibition Assays (HAI) | one month post vaccination
  Humoral immunity will be measured by hemagglutination inhibition (HAI) assay, which has been extensively used for this purpose. In healthy individuals, HAI titers ≥1:10 indicate presence of influenza-specific antibodies and ≥1:40 protection against infection and disease. In this study we will use the following definitions to assess the humoral immune response to TIV: HAI titers <1:10 = seronegative; HAI titers ≥1:10 = seropositive; HAI titers ≥1:40 = sero-protective titers; and sero-conversion will be defined as HAI titers from <1:10 to ≥1:40 or ≥4-fold increase if pre-vaccination titers were ≥1:10.

SECONDARY OUTCOMES:
impact of vaccination on T-cell activation and on T- and B-cell subpopulations | one month post vaccination
  T-lymphocyte activation assays will be performed using state-of-the art polychromatic flow cytometry. The T- and B-cell phenotypes are assessed by flow cytometry using freshly thawed Peripheral Blood Mononuclear Cells (PBMC). Cells are stained using monoclonal antibodies against the comparator molecules.
Impact of Vaccination of Cell Mediated Immune (CMI) Responses | one month post vaccination
  Interferon(IFN)Enzyme Linked Immuno Spot (ELISPOT) responses will be used to assess CMI responses to influenza vaccines.PBMCs will be separated and stimulated with influenza virus corresponding to the vaccine strains. Spots will be visualized with a ELISPOT plate reader. Results will be reported as Spot Forming Cells(SFC)/106 PBMCs.
Local and Systemic solicited reactions to TIV | 1 week and one month post vaccination
  Participants will remain in the clinic for at least 30 minutes after vaccination so that clinic personnel can observe participants for any potential adverse reactions.Report of vaccine-related local (redness, swelling, tenderness, itching,) and systemic (fever, malaise, myalgia, nausea, headache, rash) adverse events will be solicited at day 7 and day 28.
safety outcome measures of TIV | within one month post vaccination
  Safety and tolerability of the study vaccine will be monitored by means of Adverse Events (AEs) and toxicity reports presenting laboratory and clinical data.Toxicities will be classified by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events,

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, PHD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Nrf/Dst Vpd Rmpru, Soweto, Gauteng, South Africa